CLINICAL TRIAL: NCT03116087
Title: Testosterone Replacement in Postmenopausal Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Matthew Ho, Associate Professor, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5-U54-HD041748-03-D227F; 5U54HD041748-03 (NIH)
Record Dates: First submitted 2012-03-04; First posted 2017-04-14 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Postmenopausal women
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone patch (Active Comparator): Testosterone patches
  Interventions: Drug: Testosterone patch
- Placebo (Placebo Comparator): Placebo patches
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone patch — 300 mcg testosterone patches or placebo applied twice weekly
  Other Names: Testosterone patches
  Arms: Testosterone patch
Drug: Placebo — Placebo patch
  Other Names: Placebo patch
  Arms: Placebo

SUMMARY:
The overall objective of this study is to establish if testosterone replacement in post-menopausal women with low testosterone levels and stress urinary incontinence (SUI) will lead to improvement in symptoms of SUI.

This study is a prospective, randomized, double-blind, placebo-controlled, parallel-group, clinical trial and will involve sixty (60) post-menopausal women with clinically diagnosed stress urinary incontinence and low testosterone concentrations. These subjects will enter the control period, which involves the baseline measurements of pelvic floor muscle volume and strength, amounts of urine leakage in 24-hour period, urodynamic parameters, and quality of life using Incontinence Impact Questionnaire and Urogenital Distress Inventory. Subjects are then randomly assigned to either placebo (30 subjects) or 300 mcg/twice-weekly testosterone patch (30 subjects) group. Both the subjects and investigators will be blinded. The duration of the testosterone/control study will be 36 weeks, with weeks 1-3 screening/control period, 4-28 application of placebo or testosterone patches and 29-36 recovery time/assessment of effects.

DETAILED DESCRIPTION:
Primary Outcome Measure:

Our primary outcome measure is the change in levator ani muscle volume with correlation in improvement in stress incontinence. These will be assessed by MRI, urodynamic studies and pad tests. [Time Frame: 36 weeks]

Secondary Outcome Measures:

Our secondary outcome measures are: [Time Frame: 36 weeks]

1. Change in urodynamic measurements including urethral pressure profile, cough stress profile, maximum urethral closure pressure, Valsalva leak point pressure, and pressure transmission ratios.
2. Change in pelvic floor muscle strength as measured with a perineometer.
3. Change in amounts of urinary leakage (in a 24 hour period) using the Pad Test.
4. Change in subjective quality of life as it relates to incontinence using the Incontinence Impact Questionnaire, Urogenital Distress Inventory and Incontinence Diary.
5. Change in hormone levels including total and free testosterone, dihydrotestosterone (DHT), estradiol 17 B, and sex hormone binding globulin (SHBG).
6. Change in complete blood count, chem 20, lipid profile (total cholesterol, triglyceride, HDL, LDL) and physical examination as compared to the baseline before treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Ambulatory, postmenopausal women
  * The presence of stress urinary incontinence, defined as involuntary urine loss during physical activity, cough, or sneeze.
  * Able to understand and give informed consent.
  * Those on estrogen replacement therapy prior to the study should have been on a stable regimen for at least three months. For those who are not on estrogen replacement therapy prior to the study, will not be started on estrogen for the duration of the study.
  * Normal Pap smear and mammogram in the preceding 12 months by history and chart review.

Exclusion Criteria:

* Uncontrolled depression as assessed by history and physical exam.
* Those with any acute or chronic illness, malignant disease, fever of known or unknown origin, diabetes mellitus (fasting blood glucose > 126 mg/dl), or uncontrolled hypertension (defined as blood pressure greater than 160/100).
* Current urinary tract infection (UTI). For those with acute UTI, treatment will be given and repeat culture should be negative before enrollment.
* Severe obesity defined as body mass index of greater than 40 kg/m2.
* Current or recent (last 6 months) use of illicit drugs (which may affect appetite, food intake, metabolism, and/or compliance with the protocol).
* Current or recent (last 6 months) alcohol or drug dependence.
* Significant liver function abnormalities defined as AST, ALT, or alkaline phosphatase value of greater than three times the upper limit of normal in our Clinical Pathology Laboratory, or serum bilirubin levels of greater than 2 mg/dl.
* History of breast or endometrial cancer.
* History of hyperandrogenic disorders such as hirsutism and polycystic ovary disease.
* Previous intolerance to testosterone.
* Women with abnormal PAP smears or mammograms will be included only after they have been evaluated by their gynecologists and breast and uterine/cervical cancers have been excluded by appropriate diagnostic tests.
* Women with significant dementia as assessed by history and physical exam.
* Those with disabilities that would prevent them from participating in the outcome testing, including tests of pelvic floor strength (e.g. severe arthritis, Parkinson's disease, stroke, or myopathy).
* Those who have received in the preceding three months drugs known to affect testosterone production or metabolism such as Ketoconazole, Megace, and or anabolic/androgenic steroids.
* Because of their age and post-menopausal status, spontaneous pregnancy is unlikely. Regardless, women who are pregnant, seeking to become pregnant in the next six months, or breastfeeding will not be included.
* Subjects who cannot have an MRI due to metal implants or pacemaker.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Our primary outcome measure is the change in levator ani muscle volume with correlation in improvement in stress incontinence. | 36 weeks
  This outcome will be assessed by MRI, urodynamic studies and pad tests.

SECONDARY OUTCOMES:
Change in urethral pressure profile. | 36 weeks
  This outcome will be evaluated with urodynamic measurement of urethral pressure (in cm H2O) along the urethra.
Change in pelvic floor muscle strength. | 36 weeks
  This outcome will be measured with a perineometer.
Change in amounts of urinary leakage. | 36 weeks
  This will be measured with the Pad Test ( in a 24 hour period).
Change in subjective quality of life as it relates to incontinence. | 36 weeks
  This outcome will be measured with a validated questionnaire and compared with the baseline before treatment.
Change in hormone levels including total and free testosterone, dihydrotestosterone (DHT), estradiol 17 B, sex hormone binding globulin (SHBG). | 36 weeks
  These will be measured at the baseline (before treatment) and then every four weeks during the treatment and recovery periods and compared with the baseline.
Change in laboratory values. | 36 weeks
  The blood sample will be collected for laboratory measurement (CBC, chem 20, lipid profile) at the baseline (before treatment) and then every four weeks during the treatment and recovery periods and compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H Ho, MD, Principal Investigator — Charles R. Drew University
Locations (1):
- Charles R. Drew University of Medicine and Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share IPD: Presentation (grand rounds, scientific meetings) and peer-reviewed publications.